CLINICAL TRIAL: NCT02112682
Title: The Value of Completion Axillary Treatment in Sentinel Node Positive Breast Cancer Patients Undergoing a Mastectomy. A Dutch Randomized Controlled Multicentre Trial.
Brief Title: Omitting Completion Axillary Treatment in Sentinel Node Positive Breast Cancer Patients Undergoing a Mastectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual rate
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Borstkanker Onderzoek Groep (Network); Dutch Cancer Society (Other); Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BOOG 2013-07; KWF UM 2013-5920 (Other Grant/Funding Number: Dutch Cancer Society (in Dutch: KWF Kankerbestrijding))
Record Dates: First submitted 2014-04-10; First posted 2014-04-14 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Breast Neoplasms
Keywords: Sentinel lymph node metastasis; Completion axillary lymph node dissection; Axillary radiotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Completion axillary treatment (Active Comparator): Completion axillary treatment according to the Dutch breast cancer guideline
  Interventions: Procedure: Completion axillary treatment
- No completion axillary treatment (No Intervention)

INTERVENTIONS:
Procedure: Completion axillary treatment — Completion axillary treatment according to the Dutch breast cancer guideline
  Arms: Completion axillary treatment

SUMMARY:
STUDY AIM To decrease the number of breast cancer patients receiving overtreatment of the axilla, in order to positively influence the axillary morbidity rate and quality of life.

PRIMARY OBJECTIVE To determine whether omitting completion axillary treatment is not inferior to the current axillary treatment regimen in sentinel node positive breast cancer patients undergoing a mastectomy, in terms of regional recurrence rate.

HYPOTHESIS Completion axillary treatment can be safely omitted in sentinel node positive breast cancer patients undergoing a mastectomy. This will lead to a decreased axillary morbidity rate and to an increased quality of life, with non-inferior regional control, distant-disease free- and overall survival rates.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18 years or older
* Pathologically confirmed invasive unilateral breast carcinoma
* A clinical T1-2 tumour (including multifocal or multicentric breast cancer)
* Will be or is treated with mastectomy
* Clinically node negative: no signs of axillary lymph node metastases at physical examination and preoperative axillary ultrasound (or negative cyto-/histopathology)
* Sentinel lymph node procedure and its pathologic evaluation should be performed according to the Dutch breast cancer guideline
* pN1mi(sn) or pN1(sn): at least one and a maximum of three axillary sentinel lymph nodes containing micro- and/or macrometastases
* Written informed consent

Exclusion Criteria:

* Clinically node positive pre-operative
* Sentinel lymph nodes only containing isolated tumour cells (<0.2 mm)
* Solitary parasternal sentinel lymph node metastasis (pN1b)
* Bilateral breast cancer
* Irradical resection of primary tumour at time of randomization (applicable in case the mastectomy is performed before randomization)
* Evidence of metastatic disease
* History of invasive breast cancer
* Previous treatment of the axilla with surgery or radiotherapy (except surgery for hidradenitis suppurativa or for other superficially located skin lesions, such as naevi)
* Pregnant or nursing
* Other prior malignancies within the past 5 years (except successfully treated basal cell and squamous cell skin cancer, carcinoma in situ of the cervix or carcinoma in situ of the ipsilateral or contralateral breast) or unsuccessfully treated malignancies > 5 years before randomization
* Unable or unwilling to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2014-06; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Regional recurrence rate | up to ten years
  Regional recurrence is defined as tumour recurrence and as residual tumour that became clinically apparent in ipsilateral axillary, infraclavicular and supraclavicular lymph nodes (pathologically proven).

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein L Smidt, MD, PhD, Principal Investigator — Maastricht University Medical Centre+, Maastricht, the Netherlands; Hans JW de Wilt, MD, PhD, Principal Investigator — Radboud University Medical Centre, Nijmegen, the Netherlands
Locations (31):
- Netherlands (31):
  - Maastricht University Medical Centre+, Maastricht, Limburg
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Flevoziekenhuis, Almere Stad
  - Meander Medisch Centrum, Amersfoort
  - Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn
  - Rijnstate, Arnhem
  - Amphia ziekenhuis, Breda
  - Reinier de Graaf, Delft
  - Deventer Ziekenhuis, Deventer
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - UMC Groningen, Groningen
  - Zuyderland Medisch Centrum, Heerlen
  - Tergooi, Hilversum
  - Alrijne ziekenhuis, Leiden
  - St. Antonius Ziekenhuis, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Radboud university medical center, Nijmegen
  - Laurentius Ziekenhuis, Roermond
  - Zuyderland Medisch Centrum, Sittard
  - Antonius Ziekenhuis, Sneek
  - Bronovo / Medisch Centrum Haaglanden, The Hague
  - Haga Ziekenhuis, The Hague
  - Rivierenland, Tiel
  - St. Elisabeth Ziekenhuis, Tilburg
  - Diakonessenhuis Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - Isala Klinieken, Zwolle

REFERENCES:
- [Derived] van Roozendaal LM, de Wilt JH, van Dalen T, van der Hage JA, Strobbe LJ, Boersma LJ, Linn SC, Lobbes MB, Poortmans PM, Tjan-Heijnen VC, Van de Vijver KK, de Vries J, Westenberg AH, Kessels AG, Smidt ML. The value of completion axillary treatment in sentinel node positive breast cancer patients undergoing a mastectomy: a Dutch randomized controlled multicentre trial (BOOG 2013-07). BMC Cancer. 2015 Sep 3;15:610. doi: 10.1186/s12885-015-1613-2. PMID 26335105